CLINICAL TRIAL: NCT00948090
Title: A Multi-center, Phase 2, Single-Arm, Open-Label Exploratory Study of Individually- Optimized Conditioning Using Pharmacokinetics [PK]-Directed Dose Adjustment of Once Daily Intravenous Busulfan, Followed by Autologous Hematopoietic Stem Cell Transplant in Subjects With Non-Hodgkin's Lymphoma and Hodgkin's Lymphoma
Brief Title: PK-directed Dose Adjustment of IV Busulfan Conditioning Regimen for Autologous Stem Cell Transplant in Lymphoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Center for International Blood and Marrow Transplant Research (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 273-08-201
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Results first posted 2014-07-31 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Lymphoma
Keywords: Hodgkin Lymphoma; Non-Hodgkin's Lymphoma; Bone marrow transplant; stem cell transplant; busulfan; cyclophosphamide; etoposide
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Busulfan; Cyclophosphamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IV Busulfan (Experimental): Pk-directed IV Busulfan (based on test dose method) for 4 days followed by Etoposide 1400mg/m2 QD for one day and Cyclophosphamide 2.5 g/m2 QD for two days followed by autologous stem cell transplant
  Interventions: Drug: IV Busulfan, Cyclophosphamide and Etoposide (BuCyE Regimen)

INTERVENTIONS:
Drug: IV Busulfan, Cyclophosphamide and Etoposide (BuCyE Regimen) — Pk-directed IV Busulfan (based on test dose method) for 4 days followed by Etoposide 1400mg/m2 QD for one day and Cyclophosphamide 2.5 g/m2 QD for two days followed by autologous stem cell transplant.

SUMMARY:
This is a study for the outcome and safety of individualized busulfan dosing with cyclophosphamide and etoposide for patients preparing for a stem cell transplant to treat Non-Hodgkin or Hodgkin's Lymphoma.

DETAILED DESCRIPTION:
Evaluation of progression-free survival, transplant related mortality, overall survival, and overall response rate, in subjects with NHL and HL receiving an IV busulfan-based conditioning regimen with PK-guided IV busulfan dosing, followed by autologous HSCT as well as comparison to those receiving carmustine, etoposide, cytarabine, and melphalan (BEAM) conditioning regimen (and its variants) obtained from registry data in the Center for International Blood and Marrow Transplant Research (CIBMTR) Assessment of the safety profile of a BuCyE conditioning regimen with PK-directed dosing of IV busulfan will also be completed.

ELIGIBILITY:
Inclusion Criteria:

Subjects with NHL to be included:

* Any subject with NHL that had relapsed or progressed following initial therapy with an anthracycline-based chemotherapy regimen and has achieved a subsequent partial remission (PR) or a complete remission (CR) following a salvage chemotherapy regimen.
* Any subject with NHL that was initially refractory to an anthracycline-based chemotherapy regimen but who has achieved a PR or CR following a salvage chemotherapy regimen.
* Any subject with an initial International Prognostic Index (IPI) score 4-5 who achieved a PR or any CR following an anthracycline-based chemotherapy regimen except subjects with Mantle cell, T cell and Natural Killer (NK) cell pathologies.
* Subjects with Mantle cell, T cell and NK cell lymphoma may be enrolled if they have PR or CR after initial therapy.
* Any subject that has relapsed or progressed following previous autologous HSCT.

Subjects with HL to be included:

* Any subject with HL that had relapsed or progressed following initial therapy with an multi-drug chemotherapy regimen and has achieved a subsequent PR or a CR following a salvage chemotherapy regimen.
* Any subject with HL that is initially refractory to a multi-drug chemotherapy regimen but who has achieved a PR or CR following a salvage chemotherapy regimen.
* Any subject that has relapsed or progressed following previous autologous HSCT.

Exclusion Criteria:

* Any subject with chemoresistant disease by demonstration of less than PR to most recent chemotherapy, and any subject with prior treatment history of autologous HSCT or high-dose chemotherapy with stem cell rescue for any medical reason will be excluded.

Excluded will also be subjects with existing or active central nervous system lymphoma or human immunodeficiency virus related lymphoma, unacceptable organ function, or uncontrolled infections.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2010-01; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Elekes, MD, Study Director — Otsuka Pharmaceutical Development and commercialization
Locations (42):
- United States (37):
  - University of Alabama in Birmingham, Birmingham, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - Alta Bates Summit Medical Center, Berkeley, California
  - Scripps Clinic, La Jolla, California
  - UCSD Medical Center BMT Program, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Sutter Cancer Center, Sacramento, California
  - University of California, Davis Medical Center, Sacramento, California
  - University of California San Francisco Medical Center, San Francisco, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - University of Illinois Cancer Center, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - Loyola University Chicago, Maywood, Illinois
  - Bone Marrow and Stem Cell Transplant Program, Indianapolis, Indiana
  - University of Kansas Medical Center, Westwood, Kansas
  - LSU Health Sciences Center at Shreveport/Feist Weiller Cancer Center, Shreveport, Louisiana
  - University of Maryland Medical Center - Marlene & Stewart Greenebaum Cancer Center, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Weill Cornell Medical College, New York, New York
  - Montefiore-Einstein Cancer Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - The Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - South Texas Veterans Health Care System, San Antonio, Texas
  - Texas Transplant Physician Group, PLLC, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - West Virginia University Hospital, Morgantown, West Virginia
- Canada (5):
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Queen Elizabeth II Health Sciences Centre - VG Site, Halifax, Nova Scotia
  - The Ottawa Hospital, Ottawa, Ontario
  - Royal Victoria Hospital MUHC, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multicenter (43 trial sites in United States and Canada), single-arm, open-label, phase 2 exploratory trial to evaluate clinical outcomes following pharmacokinetic (PK)-directed intravenous (IV) busulfan therapy in 207 participants with Non-Hodgkin's and Hodgkin's lymphoma were evaluated.
Pre-assignment Details: Test dose of 0.8 mg/kg of IV busulfan was administered (2-hour continuous infusion) 1 day between Days -14 and -11 for PK analysis to inform subsequent dosing. The conditioning regimen consisted of IV busulfan on Days -8 to -5, etoposide on Day -4, and cyclophosphamide on Days -3 and -2, followed by stem cell infusion on Day 0.
Groups:
- Hodgkin's Lymphoma (≤ 65 Years): Participants with Hodgkins lymphoma whose age was ≤ 65 years; who received a test dose of 0.8 mg/kg of IV busulfan between Days -14 and -11; and recieved conditioning regimen of IV busulfan once daily on Days -8 to -5, etoposide on Day -4, and cyclophosphamide on Days -3 and -2, followed by stem cell infusion on Day 0.
- Hodgkin's Lymphoma (> 65 Years): Participants with Hodgkins lymphoma whose age was > 65 years; who received a test dose of 0.8 mg/kg of IV busulfan between Days -14 and -11; and recieved conditioning regimen of IV busulfan once daily on Days -8 to -5, etoposide on Day -4, and cyclophosphamide on Days -3 and -2, followed by stem cell infusion on Day 0.
- Non-Hodgkin's Lymphoma (≤ 65 Years): Participants with Non-Hodgkins lymphoma whose age was ≤ 65 years; who received a test dose of 0.8 mg/kg of IV busulfan between Days -14 and -11; and recieved conditioning regimen of IV busulfan once daily on Days -8 to -5, etoposide on Day -4, and cyclophosphamide on Days -3 and -2, followed by stem cell infusion on Day 0.
- Non-Hodgkin's Lymphoma (> 65 Years): Participants with Non-Hodgkins lymphoma whose age was > 65 years; who received a test dose of 0.8 mg/kg of IV busulfan between Days -14 and -11; and recieved conditioning regimen of IV busulfan once daily on Days -8 to -5, etoposide on Day -4, and cyclophosphamide on Days -3 and -2, followed by stem cell infusion on Day 0.
Period: Overall Study
Arm/Group | Hodgkin's Lymphoma (≤ 65 Years) | Hodgkin's Lymphoma (> 65 Years) | Non-Hodgkin's Lymphoma (≤ 65 Years) | Non-Hodgkin's Lymphoma (> 65 Years)
Started | 65 | 1 | 123 | 18
Completed | 22 | 0 | 67 | 7
Not Completed | 43 | 1 | 56 | 11

BASELINE CHARACTERISTICS:
Groups:
- Hodgkin's/Non-Hodgkin's Lymphoma (≤ 65 Years): Participants with Hodgkin's or Non-Hodgkins lymphoma whose age was ≤ 65 years; who received a test dose of 0.8 mg/kg of IV busulfan between Days -14 and -11; and recieved conditioning regimen of IV busulfan once daily on Days -8 to -5, etoposide on Day -4, and cyclophosphamide on Days -3 and -2, followed by stem cell infusion on Day 0.
- Hodgkin's/Non-Hodgkin's Lymphoma (> 65 Years): Participants with Hodgkin's or Non-Hodgkins lymphoma whose age was > 65 years; who received a test dose of 0.8 mg/kg of IV busulfan between Days -14 and -11; and recieved conditioning regimen of IV busulfan once daily on Days -8 to -5, etoposide on Day -4, and cyclophosphamide on Days -3 and -2, followed by stem cell infusion on Day 0.
- Total: Total of all reporting groups
Arm/Group | Hodgkin's/Non-Hodgkin's Lymphoma (≤ 65 Years) | Hodgkin's/Non-Hodgkin's Lymphoma (> 65 Years) | Total
Number analyzed (Participants) | 188 | 19 | 207
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Years | 46.5 (13.1) | 68.5 (2.3) | 48.5 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 2 | 68
  Male | 122 | 17 | 139

OUTCOME MEASURES:

1. Primary Outcome: Number of Progression Events in 2 Years.
Description: The time of Progression-Free Survival (PFS) was defined as the time from transplantation to the occurrence of the event that was death or first recurrence of progressive disease.
Time Frame: 2 years
Population: Participants receiving at least 1 PK-directed IV busulfan dose followed by autologous hematopoietic stem cell transplant are included in the Intent-to-treat (ITT) data set. Four participants (of 207) did not continue to the conditioning regimen after receiving the PK test dose and were excluded from ITT data set.
Measure: Number; unit: Event
Arm/Group | Hodgkin's Lymphoma (≤ 65 Years) | Hodgkin's Lymphoma (> 65 Years) | Non-Hodgkin's Lymphoma (≤ 65 Years) | Non-Hodgkin's Lymphoma (> 65 Years)
Number analyzed (Participants) | 65 | 1 | 121 | 16
Event | 41 | 1 | 46 | 8

2. Secondary Outcome: Number of Death Events in 2 Years.
Description: The time of overall survival was defined as the time from transplantation to death of all causes.
Time Frame: 2 years
Population: Participants receiving at least 1 PK-directed IV busulfan dose followed by autologous hematopoietic stem cell transplant are included in the ITT data set. Four participants (of 207) did not continue to the conditioning regimen after receiving the PK test dose and were excluded from ITT data set.
Measure: Number; unit: Deaths
Arm/Group | Hodgkin's Lymphoma (≤ 65 Years) | Hodgkin's Lymphoma (> 65 Years) | Non-Hodgkin's Lymphoma (≤ 65 Years) | Non-Hodgkin's Lymphoma (> 65 Years)
Number analyzed (Participants) | 65 | 1 | 121 | 16
Deaths | 13 | 1 | 28 | 6

3. Secondary Outcome: Number of Transplant-related Death Events Until Day 100.
Description: Transplant-related mortality was defined as death due to any cause other than disease relapse/progression up until Day 100.
Time Frame: Day 100
Population: as for outcome 2
Measure: Number; unit: Transplant-related death
Arm/Group | Hodgkin's Lymphoma (≤ 65 Years) | Hodgkin's Lymphoma (> 65 Years) | Non-Hodgkin's Lymphoma (≤ 65 Years) | Non-Hodgkin's Lymphoma (> 65 Years)
Number analyzed (Participants) | 65 | 1 | 121 | 16
Transplant-related death | 1 | 1 | 5 | 3

4. Secondary Outcome: Overall Response Rate
Description: The overall response status is complete response and not complete response (partial remission, primary refractory/primary induction failure, stable disease, progressive disease, and relapse) at Baseline and each of the scheduled follow-up time points.
Time Frame: Baseline, Day 100, Month 6, 12, 24, Early termination and End of Trial (within 30 days of the trial termination)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Hodgkin's Lymphoma (≤ 65 Years) | Hodgkin's Lymphoma (> 65 Years) | Non-Hodgkin's Lymphoma (≤ 65 Years) | Non-Hodgkin's Lymphoma (> 65 Years)
Number analyzed (Participants) | 65 | 1 | 121 | 16
Participants
  Baseline-Complete Response (N=65, 0, 121, 16) | 35 | 0 | 72 | 12
  Baseline-Not Complete Response (N=65, 1, 121, 16) | 30 | 1 | 49 | 4
  Day 100-Complete Response (N=57, 0, 114, 12) | 35 | 0 | 85 | 8
  Day 100-Not Complete Response (N=57, 0, 114, 12) | 22 | 0 | 29 | 4
  Month 6-Complete Response (N=45, 0, 98, 11) | 30 | 0 | 84 | 9
  Month 6-Not Complete Response (N=45, 0, 98, 11) | 15 | 0 | 14 | 2
  Month 12-Complete Response (N=32, 0, 88, 8) | 22 | 0 | 71 | 8
  Month 12-Not Complete Response (N=32, 0, 88, 0) | 10 | 0 | 17 | 0
  Month 24-Complete Response (N=13, 0, 28, 6) | 11 | 0 | 26 | 6
  Month 24-Not Complete Response (N=13, 0, 28, 0) | 2 | 0 | 2 | 0
  Early Term-Complete Response (N=40, 0, 41, 0) | 2 | 0 | 4 | 0
  Early Term-Not Complete Response (N=40, 0, 41, 5) | 38 | 0 | 37 | 5
  End of Trial-Complete Response (N=22, 0, 71, 9) | 20 | 0 | 65 | 8
  End of Trial-Not Complete Response(N=22, 0, 71, 9) | 2 | 0 | 6 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were reported during the entire trial period (from screening through Early Termination or End of Trial).
Groups:
- Hodgkin's/Non-Hodgkin's Lymphoma (≤ 65 Years or > 65 Years): The safety data set consisted of all screened participants who had received at least 1 dose of IV busulfan (including PK test dose).
Arm/Group | Hodgkin's/Non-Hodgkin's Lymphoma (≤ 65 Years or > 65 Years)
Serious Adverse Events (participants affected / at risk) | 90/207
Other Adverse Events (participants affected / at risk) | 190/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hodgkin's/Non-Hodgkin's Lymphoma (≤ 65 Years or > 65 Years) (N=207)
Anaemia (Blood and lymphatic system disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 9
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Atrial fibrillation (Cardiac disorders) | 5
Atrial thrombosis (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardiac tamponade (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Diabetes insipidus (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Gastrointestinal toxicity (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 1
Multi-organ failure (General disorders) | 2
Pyrexia (General disorders) | 9
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholecystits chronic (Hepatobiliary disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1
Hepatic vein occlusion (Hepatobiliary disorders) | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 1
Cytokine storm (Immune system disorders) | 1
Acinetobacter bacteraemia (Infections and infestations) | 1
Aspergillosis (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 2
Bacterial infection (Infections and infestations) | 2
Bacterial sepsis (Infections and infestations) | 1
BK virus infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Clostridial infection (Infections and infestations) | 1
Clostridium Difficile colitis (Infections and infestations) | 1
Cystitis viral (Infections and infestations) | 1
Cytomegalovirus viraemia (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lung infection (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 9
Pneumonia fungal (Infections and infestations) | 1
Pneumonia pneumococcal (Infections and infestations) | 1
Pulmonary mycosis (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 1
Salmonella bacteraemia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 8
Septic shock (Infections and infestations) | 4
Staphylococcal infection (Infections and infestations) | 1
Syphilis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection Enterococcal (Infections and infestations) | 1
Viraemia (Infections and infestations) | 1
Delayed engraftment (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1
Blood culture positive (Investigations) | 1
Pulmonary physical examination abnormal (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Failure to thrive (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
IIIrd nerve paralysis (Nervous system disorders) | 1
Vocal cord paralysis (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Renal failure acute (Renal and urinary disorders) | 6
Renal tubular necrosis (Renal and urinary disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pleural haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 7
Hypovolaemic shock (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Hodgkin's/Non-Hodgkin's Lymphoma (≤ 65 Years or > 65 Years) (N=207)
Anaemia (Blood and lymphatic system disorders) | 22
Febrile neutropenia (Blood and lymphatic system disorders) | 129
Neutropenia (Blood and lymphatic system disorders) | 23
Thrombocytopenia (Blood and lymphatic system disorders) | 27
Atrial fibrillation (Cardiac disorders) | 12
Sinus tachycardia (Cardiac disorders) | 12
Tachycardia (Cardiac disorders) | 39
Dry eye (Eye disorders) | 12
Abdominal distension (Gastrointestinal disorders) | 19
Abdominal pain (Gastrointestinal disorders) | 61
Abdominal pain upper (Gastrointestinal disorders) | 14
Constipation (Gastrointestinal disorders) | 70
Diarrhoea (Gastrointestinal disorders) | 179
Dry mouth (Gastrointestinal disorders) | 30
Dyspepsia (Gastrointestinal disorders) | 46
Dysphagia (Gastrointestinal disorders) | 19
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 19
Haemorrhoids (Gastrointestinal disorders) | 37
Nausea (Gastrointestinal disorders) | 169
Oesophagitis (Gastrointestinal disorders) | 18
Oral pain (Gastrointestinal disorders) | 23
Proctalgia (Gastrointestinal disorders) | 19
Stomatitis (Gastrointestinal disorders) | 170
Vomiting (Gastrointestinal disorders) | 132
Asthenia (General disorders) | 28
Catheter site erythema (General disorders) | 12
Chest discomfort (General disorders) | 12
Chest pain (General disorders) | 18
Chills (General disorders) | 38
Fatigue (General disorders) | 104
Mucosal inflammation (General disorders) | 11
Oedema (General disorders) | 20
Oedema peripheral (General disorders) | 68
Pain (General disorders) | 31
Pyrexia (General disorders) | 94
Hyperbilirubinaemia (Hepatobiliary disorders) | 19
Oral candidiasis (Infections and infestations) | 13
Pneumonia (Infections and infestations) | 12
Upper respiratory tract infection (Infections and infestations) | 21
Excoriation (Injury, poisoning and procedural complications) | 11
Alanine aminotransferase increased (Investigations) | 25
Aspartate aminotransferase increased (Investigations) | 29
Blood alkaline phosphatase increased (Investigations) | 18
Blood bilirubin increased (Investigations) | 13
Blood creatinine increased (Investigations) | 15
Gamma-glutamyltransferase increased (Investigations) | 11
Haemoglobin decreased (Investigations) | 13
Platelet count decreased (Investigations) | 19
Weight decreased (Investigations) | 32
White blood cell count decreased (Investigations) | 19
Decreased appetite (Metabolism and nutrition disorders) | 94
Dehydration (Metabolism and nutrition disorders) | 13
Fluid overload (Metabolism and nutrition disorders) | 22
Hyperglycaemia (Metabolism and nutrition disorders) | 26
Hypoalbuminaemia (Metabolism and nutrition disorders) | 23
Hypocalcaemia (Metabolism and nutrition disorders) | 26
Hypokalaemia (Metabolism and nutrition disorders) | 100
Hypomagnesaemia (Metabolism and nutrition disorders) | 63
Hyponatraemia (Metabolism and nutrition disorders) | 36
Hypophosphataemia (Metabolism and nutrition disorders) | 48
Arthralgia (Musculoskeletal and connective tissue disorders) | 13
Back pain (Musculoskeletal and connective tissue disorders) | 22
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18
Dizziness (Nervous system disorders) | 42
Dysguesia (Nervous system disorders) | 39
Headache (Nervous system disorders) | 73
Neuropathy peripheral (Nervous system disorders) | 16
Anxiety (Psychiatric disorders) | 51
Confusional state (Psychiatric disorders) | 17
Depression (Psychiatric disorders) | 21
Hallucination (Psychiatric disorders) | 16
Insomnia (Psychiatric disorders) | 86
Dysuria (Renal and urinary disorders) | 19
Haematuria (Renal and urinary disorders) | 15
Urinary retention (Renal and urinary disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 64
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 46
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 43
Hiccups (Respiratory, thoracic and mediastinal disorders) | 17
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 17
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 20
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 31
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 14
Productive cough (Respiratory, thoracic and mediastinal disorders) | 12
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 17
Wheezing (Respiratory, thoracic and mediastinal disorders) | 11
Alopecia (Skin and subcutaneous tissue disorders) | 19
Dry skin (Skin and subcutaneous tissue disorders) | 14
Erythema (Skin and subcutaneous tissue disorders) | 36
Night sweats (Skin and subcutaneous tissue disorders) | 14
Pruritis (Skin and subcutaneous tissue disorders) | 27
Rash (Skin and subcutaneous tissue disorders) | 70
Skin exfoliation (Skin and subcutaneous tissue disorders) | 12
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 15
Flushing (Vascular disorders) | 15
Hypertension (Vascular disorders) | 17
Hypotension (Vascular disorders) | 52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No